CLINICAL TRIAL: NCT02736383
Title: Effectiveness of Tranexamic Acid (TXA) in Reducing Blood Loss in Hip Fracture Surgery
Brief Title: Tranexamic Acid in Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-060
Record Dates: First submitted 2016-03-29; First posted 2016-04-13 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tranexamic Acid: Patients that receive 2 gm TXA during surgery
- No Tranexamic Acid: Patients that receive no TXA during surgery

SUMMARY:
To determine if TXA utilization is effective at reducing transfusion rates in elderly patients undergoing surgery for treatment of a hip fractures.

ELIGIBILITY:
Inclusion Criteria:

* Acute, isolated, unilateral femoral neck, intertrochanteric, and per trochanteric hip fractures confirmed by anteroposterior/lateral hip radiographs, computed tomography, or magnetic resonance imaging.
* Age 65 and older
* Low energy mechanism of injury
* Hip fracture fixation performed within 48 hours
* English speaking
* Anticipated medical optimization for operative fixation
* No other major trauma

Exclusion Criteria:

* Retained hardware around the affected hip
* Infection around the affected hip
* Transfer patients with a length of stay > 24 hours at the transferring hospital
* Diagnosis of deficient natural anticoagulation
* Known congenital thrombophilia (Deficiency of Protein C, S, Antithrombin)
* Known allergy to TXA
* Patients undergoing percutaneous pinning of the hip fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with hip fractures
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Blood Transfusion Rate | 6 weeks
  Blood transfusion rates during the patients hospital stay will be assessed.

SECONDARY OUTCOMES:
Hospital Length of stay | 6 weeks
  The patients length of stay in the hospital will be determined.
Post operative complications | 6 weeks
  Post operative complications will be assessed through the 6 weeks.
Hospitalization costs | 6 weeks
  Economic evaluation for inpatient and re-admission will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Blake W Miller, DO, Principal Investigator — Corewell Health West

IPD SHARING:
Plan to Share IPD: No